CLINICAL TRIAL: NCT00204464
Title: Preliminary Study: The Effects of a Strengthening Program on Maximum Voluntary Isometric Contraction, Functional Abilities, Fatigue and Quality of Life in Individuals With Amyotrophic Lateral Sclerosis
Brief Title: Study of the Effects Strengthening Exercises in Individuals With ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Washington University School of Medicine (Other); Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALS_EX; ALSA-CM Grant
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2005-11-04 (Estimated); Status verified 2004-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Exercise
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Activity | interventions — Exercise

INTERVENTIONS:
Procedure: Exercise

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is the most common motor neuron disease MND) among adults. Motor neurons in the spinal cord, brain stem, and cerebral motor cortex degenerate and create a variety of upper (UMN) and lower motor neuron (LMN) clinical signs and symptoms, with the most frequently presenting symptom being focal weakness beginning in the leg, arm, or bulbar muscles, occurring in more than 70% of patients. Despite the high incidence of muscle weakness in patients with ALS, only two case studies evaluating the effects of specific muscle strengthening and endurance exercise programs in this patient population have been published, and the effects of resistive exercise programs in patients with ALS have not been well studied. Some have discouraged exercise programs in patients with ALS because of fear of overuse weakness. Yet, in patients with other neuromuscular diseases, resistive exercise programs have been shown to be beneficial and have not produced overuse weakness. The purpose of this study is to determine the effects of six months strengthening program on strength, function, fatigue and quality of life in individuals with ALS.

DETAILED DESCRIPTION:
The specific aims of this preliminary, prospective randomized study of individuals with ALS are to determine variability, describe trends over a 6-month time frame and to estimate differences between individuals with ALS who perform an upper and lower extremity strengthening program three times per week and a control group of individuals with ALS with respect to the following outcomes:

1. an increase in muscle strength (maximum voluntary isometric contraction) as measured by quantitative muscle testing.
2. an increase in functional activities as measured by The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS)7 and the Schwab and England Rating Scale (SERS).
3. a decrease in fatigue as measured by the Fatigue Severity Scale.
4. an increase in quality of life as measured by the SF-36.Subjects will be randomized into two groups - experimental and control. Subjects in the control group will perform a daily stretching exercise program for a period of six months. Subjects in the experimental groups will perform a strengthening exercise program three times per week for a period of six months. All subjects will be evaluated at baseline and then monthly using the following outcome measures: (1) maximum voluntary isometric contraction; (2) Amyotrophic Lateral Sclerosis Functional Rating Scale; (3) Schwab and England Rating Scale; (3) Fatigue Severity Scale; (4) forced vital capacity; and, (5) the SF-36.

ELIGIBILITY:
Inclusion Criteria:

* definite and/or probable diagnosis of ALS
* early stages of the disease

Exclusion Criteria:

* history of neuromuscular dysfunction not related to ALS
* active, confounding medical conditions
* unwillingness or inability to comply with the protocol
* FVC of less than 90% predicted
* ALSFRS score of less than 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Study Completion 2004-12

PRIMARY OUTCOMES:
Function - ALSFRS

SECONDARY OUTCOMES:
MVIC
FVC
Fatigue
SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Vanina PM Dal Bello-Haas, PhD, BScPT, Principal Investigator — University of Saskatchewan
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States